CLINICAL TRIAL: NCT02193594
Title: Phase Ⅱ/Ⅲ Study of Preoperative Concurrent Chemoradiotherapy for Locally Advanced Gastroesophageal Junction or Upper Gastric Adenocarcinoma
Brief Title: Preoperative Concurrent Chemoradiotherapy for Locally Advanced Gastroesophageal Junction or Upper Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Chinese PLA General Hospital (Other); Peking University People's Hospital (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jiafu Ji, President of Beijing Cancer Hospital,Director of Key Laboratory of Carcinogenesis and Translational Research(Gastric Cancer Laboratory), Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRADLE
Record Dates: First submitted 2014-07-08; First posted 2014-07-17 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Gastroesophageal Junction Adenocarcinoma
Keywords: Preoperative concurrent chemoradiotherapy; Neoadjuvant chemoradiotherapy; Gastroesophageal junction adenocarcinoma
MeSH Terms: interventions — Oxaliplatin; S 1 (combination); Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CCRT group (Experimental): The patient in CCRT group will receive the preoperative concurrent chemoradiotherapy for 5 weeks and sequential radical D2 total gastrectomy and postoperative adjuvant chemotherapy of 6 cycles.
  Interventions: Radiation: Preoperative concurrent chemoradiotherapy; Procedure: Radical D2 total gastrectomy; Drug: Adjuvant chemotherapy
- CT group (Active Comparator): The patient in CT group will receive radical D2 total gastrectomy and postoperative adjuvant chemotherapy of 8 cycles.
  Interventions: Procedure: Radical D2 total gastrectomy; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Radiation: Preoperative concurrent chemoradiotherapy — The patients will receive radiotherapy in the total amount of 50Gy(25 fractions) preoperatively,concurrently combined with chemotherapy,which consist of oxaliplatin 40mg/m2 administrated on days 1,8,15,22,29 and S-1® 30mg/m2 twice per day on days 1 to 5 per week.
  Other Names: CCRT; Eloxatin®; S-1®
  Arms: CCRT group
Procedure: Radical D2 total gastrectomy — Within 5-6 weeks after the completion of neoadjuvant therapy,the patients in CCRT group will receive the radical total gastrectomy with D2 lymphadenectomy,and patients in the CT group will receive the surgery right after randomization.
Drug: Adjuvant chemotherapy — Within 2 months after surgery,the patients will receive chemotherapy for 6 to 8 cycles ,consist of oxaliplatin 130mg/m2 administrated on day1 and S-1® 40-60mg twice per day on days 1 to 14 per 3 weeks.The S-1® dosage depends on the patient BSA(BSA<1.25m2 40mg,1.25 m2≤BSA≤1.5 m2 50mg ,BSA>1.5 m2 60mg). Patients in the CCRT group will receive 6 cycles of chemotherapy and patients in the CT group will receive 8 cycles of chemotherapy.
  Other Names: Eloxatin®; S-1®

SUMMARY:
Preoperative chemoradiotherapy(CRT) had been introduced in the comprehensive treatment of gastroesophageal junction and upper gastric cancers in the decade.According to some researches,CRT had shown its good curative effects in local control and prolonged overall survival.However,the optimization scheme for CRT and its influence to surgery remains controversial.Meanwhile,there were many design flaws in the past few research,such as the lack of adjuvant chemotherapy,the insufficiency in lymphnodes dissection.We decided to carry out the trial,eliminating all the bias as far as we can,to illustrate the efficacy and safety of CRT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the gastroesophageal junction.
* Clinical stage diagnosed by endoscopic ultrasound(EUS) or computed tomography(CT) as T3-4NxM0 tumors,according to American Joint Committee on Cancer (AJCC) 7th edition.
* Eastern Cooperative Oncology Group (ECOG) performance status≤2.
* Informed consent obtained.

Exclusion Criteria:

* Combined with other malignant tumors.
* Eastern Cooperative Oncology Group (ECOG) performance status>2.
* Combined with severe organ dysfunction.
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-09 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
The patient's survival time and recurrence time | Up to 3 years
  3-year overall survival
  1-year and 3-year recurrence free survival

SECONDARY OUTCOMES:
The number of patients with complications | Within 30 days after the day of operation
  the morbidity and mortality rates within 30 days after the day of operation

OTHER OUTCOMES:
The pathologic profiles and the pathologic response rates | Within 30 days after the day of operation
  the pathologic profiles and the pathologic response rates

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Haidian District, Beijing Municipality, China